CLINICAL TRIAL: NCT01507259
Title: A Randomised Trial of Effect of Chocolate Upon Cerebrovascular Reactivity in Healthy Adult Volunteers
Brief Title: Chocolate's Effect on the Cerebral Vasculature
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Steven Burke, Sponsor's representative, NHS Greater Glasgow and Clyde
Other Study IDs: GN11MT497
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Cerebral Vasculature
Keywords: Determine effect on cerebral vasculature
MeSH Terms: interventions — Chocolate

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 100 g containing 70% or 34% cocoa: Healthy controls
  Interventions: Other: cocoa

INTERVENTIONS:
Other: cocoa — 70% versus 34%

SUMMARY:
The popularity of chocolate can largely be attributed to its mood elevating properties, research shows that it contains antioxidants that also provide physical health benefits. Dark chocolate, in particular, contains high levels of an antioxidant called epicatechin, which is known to cause changes in blood vessels by relaxing them and increasing blood flow.

Little is know about the immediate effects of chocolate consumption, or the differences between milk and dark chocolate with regards to these effects. The project will investigate the effect of a single bar of dark or milk chocolate upon blood flow to the brain, using simple ultrasound tests.

ELIGIBILITY:
Inclusion Criteria:

* No regular medication including vitamins/antioxidants
* Able to provide informed consent

Exclusion Criteria:

* Inability to perform breath-hold test
* Any known cardiovascular disease, diabetes, throid disease, high blood pressure, hyperlipidaemia or pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-02; Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Infirmary, Glasgow, United Kingdom